CLINICAL TRIAL: NCT02646865
Title: A Randomized Controlled Trial on the Efficacy of Self-Compassion Enhanced CBT vs. Standard CBT for Social Anxiety
Brief Title: Self-Compassion Enhanced CBT vs. Standard CBT for Social Anxiety (SCE-CBT)
Acronym: SCE-CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Responsible Party: Principal Investigator, Diana-Mirela Candea, PhD Candidate, Babes-Bolyai University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UBB-CLINPSY-2016-1
Record Dates: First submitted 2015-12-30; First posted 2016-01-06 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Social Anxiety Disorder
Keywords: social phobia; compassion; shame
MeSH Terms: conditions — Phobia, Social | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-Compassion Enhanced Cognitive-Behavioral Therapy (Experimental): Group Cognitive-Behavioral Therapy for social anxiety enhanced with exercises targeting self-compassion
  Interventions: Behavioral: Self-Compassion Enhanced Cognitive-Behavioral Therapy
- Cognitive-Behavioral Therapy (Active Comparator): Standard Group Cognitive-Behavioral Therapy for social anxiety
  Interventions: Behavioral: Cognitive-Behavioral Therapy

INTERVENTIONS:
Behavioral: Self-Compassion Enhanced Cognitive-Behavioral Therapy — 12 group sessions of CBT for social anxiety based on Heimberg & Becker's (2002) protocol with additional self-compassion exercises integrated into the treatment
  Arms: Self-Compassion Enhanced Cognitive-Behavioral Therapy
Behavioral: Cognitive-Behavioral Therapy — 12 group sessions of CBT for social anxiety based on Heimberg & Becker's (2002) protocol
  Arms: Cognitive-Behavioral Therapy

SUMMARY:
This study evaluates the addition of a self-compassion training in the treatment of social anxiety disorder. Half of the participants will receive a self-compassion enhanced group cognitive-behavioral therapy, while the other half will receive standard group cognitive-behavioral therapy.

DETAILED DESCRIPTION:
There is growing evidence showing that shame is associated with social anxiety. Also, empirical data shows that individuals with social anxiety have higher levels of shame compared with healthy individuals and that shame might play an important role in the maintenance of social anxiety symptoms. Although cognitive-behavioral therapy for social anxiety seems to reduce the level of shame-proneness, the magnitude of this reduction is a small one.

The purpose of this study is to test whether adding a self-compassion component (which seems to be effective in reducing shame feelings) to a cognitive-behavioral protocol would increase the efficacy of the treatment in reducing both shame-proneness and social anxiety symptoms compared with a standard cognitive-behavioral intervention.

ELIGIBILITY:
Inclusion Criteria:

* subjects diagnosed with Social Anxiety Disorders using the DSM-5 criteria
* subjects that have SAD as the primary diagnosis according to DSM-5 criteria
* exceed the cutoff scores on SPIN, SIAS, and LSAS-SR

Exclusion Criteria:

* subjects that score over 29 points at BDI-II
* display suicidal ideation (i.e., exceed a score of 2 on the suicide item of BDI-II)
* undergo other forms of treatment for SAD
* have a diagnosis of psychosis, bipolar disorder or personality disorders according to DSM-5 criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Changes in social anxiety symptoms using (Liebowitz Social Anxiety Scale; Leibowitz, 1987) | (1) baseline; (2) weekly for 11 weeks starting with the second week of treatment (2) at the of end of treatment (12 weeks after the start of the treatment) ; (3) 6 months after the end of treatment
  Self-reported measure of social anxiety symptoms
Changes in social anxiety symptoms using SPIN (Social Phobia Inventory; Connor et al., 2000) | (1) baseline; (2) after 6 weeks from the start of the treatment; (2) at the of end of treatment (12 weeks after the start of the treatment); (3) 6 months after the end of treatment
  Self-reported measure of social anxiety symptoms
Changes in social anxiety symptoms using SIAS (Social Interaction Anxiety Scale; Mattick & Clarke, 1998) | (1) baseline; (2) after 6 weeks from the start of the treatment; (2) at the of end of treatment (12 weeks after the start of the treatment); (3) 6 months after the end of treatment
  Self-reported measure of social anxiety symptoms
Changes in shame-proneness using TOSCA-3 (Test of Self-Conscious Affect-3; Tangney, Dearing, Wagner, & Gramzow, 2000) | (1) baseline; (2) after 3, 6, 9 weeks from the start of the treatment; (2) at the of end of treatment (12 weeks after the start of the treatment); (3) 6 months after the end of the treatment
  Self-reported measure of predisposition to experience shame
Changes in social anxiety disorder clinical status | at the end of the therapy
  DSM-5 semi-structured interview for social anxiety disorder

SECONDARY OUTCOMES:
Changes in self-compassion using SCS (Self-Compassion Scale; Neff, 2003) | (1) baseline; (2) after 6 weeks from the start of the treatment; (2)at the of end of treatment (12 weeks after the start of the treatment); (3) 6 months after the end of treatment
  Self-reported measure of self-compassion
Changes in self-compassion using SCSs (Self-Compassion Scale Short Form; Raes et al., 2011) | (1) baseline; (2) weekly for 11 weeks starting with the second week of treatment (2) at the of end of treatment (12 weeks after the start of the treatment); (3) 6 months after the end of treatment
  Self-reported measure of self-compassion
Changes in depressive symptoms using BDI-II (Beck Depression Inventory-II; Beck, 1996) | (1) baseline; (2) after 6 weeks from the start of the treatment; (2) at the of end of treatment (12 weeks after the start of the treatment); (3) 6 months after the end of treatment
  Self-reported measure of depressive symptoms
Changes in positive and negative affect using PANAS (Positive and Negative Affect Schedule; Watson & Clark, 1999) | (1) baseline; (2) weekly for 11 weeks starting with the second week of treatment (2) at the of end of treatment (12 weeks after the start of the treatment); (3) 6 months after the end of treatment
  Self-reported measure of positive and negative affect
Changes in positive and negative emotions using PDA (Profile of Affective Distress; Opriș & Macavei, 2005) | (1) baseline; (2) after 6 weeks from the start of the treatment; (2) at the of end of treatment (12 weeks after the start of the treatment); (3) 6 months after the end of treatment
  Self-reported measure of positive and negative emotions
Changes in irrational and rational thinking using ABS-II (Attitudes and Beliefs Scale- 2; DiGiuseppe, Leaf, Exner, & Robin, 1988) | (1) baseline; (2) after 6 weeks from the start of the treatment; (2) at the of end of treatment (12 weeks after the start of the treatment); (3) 6 months after the end of treatment
  Self-reported measure of rational and irrational beliefs
Changes in emotion regulation using ERQ (Emotion Regulation Questionnaire; Gross & John, 2003) | (1) baseline; (2) after 6 weeks from the start of the treatment; (2) at the of end of treatment (12 weeks after the start of the treatment); (3) 6 months after the end of treatment
  Self-reported measure of the use of suppression and reappraisal
Changes in emotion regulation using DERS (Difficulties in Emotion Regulation Scale; Gratz & Roemer, 2004) | (1) baseline; (2) after 6 weeks from the start of the treatment; (2) at the of end of treatment (12 weeks after the start of the treatment); (3) 6 months after the end of treatment
  Self-reported measure on emotion regulation strategies
Changes in rational and irrational beliefs using GABS (General Attitudes and Beliefs Scale; Bernard, 1998) | (1) baseline; (2) after 6 weeks from the start of the treatment; (2) at the of end of treatment (12 weeks after the start of the treatment); (3) 6 months after the end of treatment
  Self-reported measure of rational and irrational beliefs
Changes in social phobia related thoughts using BFNE (Brief Fear of Negative Evaluation Scale; Leary, 1983) | (1) baseline; (2) weekly for 11 weeks starting with the second week of treatment (2) at the of end of treatment (12 weeks after the start of the treatment); (3) 6 months after the end of treatment
  Self-reported measure of social phobia relevant negative thoughts
Changes in shame with PFQ-2 (Personal Feelings Questionnaire-2; Harder & Zalma, 1990) | (1) baseline; (2) weekly for 11 weeks starting with the second week of treatment (2) at the of end of treatment (12 weeks after the start of the treatment); (3) 6 months after the end of treatment
  Self-reported measure of shame

CONTACTS AND LOCATIONS:
Locations (1):
- Babes-Bolyai University, Cluj-Napoca, Cluj, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gilbert, P, Miles, JNV.Sensitivity to social put-down: Its relationship to perceptions of social rank, shame, social anxiety, depression, anger and self-other blame. Personality and Individual Differences, 29: 757-774, 2000.
- [Background] Gilbert, P.The relationship of shame, social anxiety and depression: The role of the evaluation of social rank. Clin Psychol Psychother, 7: 174-189, 2000.
- [Background] Fergus TA, Valentiner DP, McGrath PB, Jencius S. Shame- and guilt-proneness: relationships with anxiety disorder symptoms in a clinical sample. J Anxiety Disord. 2010 Dec;24(8):811-5. doi: 10.1016/j.janxdis.2010.06.002. Epub 2010 Jun 11. PMID 20591613
- [Background] Hedman E, Strom P, Stunkel A, Mortberg E. Shame and guilt in social anxiety disorder: effects of cognitive behavior therapy and association with social anxiety and depressive symptoms. PLoS One. 2013 Apr 19;8(4):e61713. doi: 10.1371/journal.pone.0061713. Print 2013. PMID 23620782
- [Background] Gilbert, P, Procter, S. Compassionate mind training for people with high shame and self-criticism: Overview and pilot study of a group therapy approach. Clinical Psychology and Psychotherapy, 13(6): 353-379, 2006.
- [Background] Heimberg, RG, & Becker, RE. Cognitive-behavioral group therapy for social phobia: Basic mechanisms and clinical strategies. Guilford Press, 2002.
- [Background] Lutwak, N, Ferrari, JR.. Shame-related social anxiety: Replicating a link with various social interaction measures. Anxiety, stress, and coping, 10(4): 335-34, 1997.